CLINICAL TRIAL: NCT03111459
Title: Endograft Repair of Thoracoabdominal Aortic Aneurysms (TAAA)
Brief Title: Repair of Thoracoabdominal Aortic Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christ Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Geoffrey Answini, Dr., The Christ Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISR-2016-10790
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Thoracoabdominal Aneurysm
Keywords: endograft repair,

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Study Arm (Experimental): Patients meeting primary inclusion/exclusion criteria will be enrolled in this arm and treated with the Medtronic Valiant Thoracoabdominal Stent Graft System.
  Interventions: Device: Medtronic Valiant Thoracoabdominal Stent Graft System
- Expanded Selection Arm (Experimental): Patients who fail to meet the inclusion criteria of the Primary Study Arm may be enrolled under the Expanded Selection Arm and be treated with the Medtronic Valiant Thoracoabdominal Stent Graft System.
  Interventions: Device: Medtronic Valiant Thoracoabdominal Stent Graft System

INTERVENTIONS:
Device: Medtronic Valiant Thoracoabdominal Stent Graft System — The Medtronic Valiant Thoracoabdominal Stent Graft System is made up of two main body components and makes use of several off-the-shelf FDA-approved stent graft components The system is comprised of two investigational devices that include the thoracic bifurcation and the visceral manifold. The thoracic bifurcation is deployed in the thoracic aorta and provides the proximal seal for the device. The two limbs of the thoracic bifurcation allows for continued aortic flow while deploying the visceral segment. The visceral manifold is deployed within the larger 20 mm limb of the thoracic bifurcation to set the stage for the visceral debranching. The branches of the visceral manifold extend to the visceral vessel with the use of covered bridging stents and provide distal seal of the manifold.

SUMMARY:
The primary objective of the clinical investigation is to assess the use of the Medtronic Valiant Thoracoabdominal Stent Graft System to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety and preliminary effectiveness of the device. Additionally, the study will assess technical success and treatment success at each follow-up interval.

DETAILED DESCRIPTION:
Patients diagnosed with TAAA have a poor medical history and require surgical intervention to extend life. Several repair techniques have been developed, but each carry risk. Open repairs are durable but have substantial perioperative mortality and postoperative morbidity. Endovascular techniques are plagued by high procedural complexity and poor branch vessel patency. Parallel techniques may have poor seal and may be prone to endoleak. In contrast, the manifold approach has circumferential seal at the proximal end of the system. It has relatively simple case planning and it has virtually no ischemic time. Due to these advantages, the Investigator believes the novel proposed technique may overcome some of the current clinical risks with other approaches.

Patients who participate in this study may benefit from having a less invasive procedure compared to open repair of their thoracoabdominal aortic aneurysm. The Investigator expects the amount of discomfort, total blood loss, recovery time, and overall hospital stay to be less than open repair. Many of the patients presenting with a thoracoabdominal aneurysm are not candidates for open repair due to existing comorbidities. With the progressive nature of the disease, these patients have limited options for medical intervention and are willing to assume a higher amount of risk.

The Medtronic Valiant Thoracoabdominal Stent Graft System is made up of two main body components and makes use of several off-the-shelf FDA-approved stent graft components. The two custom main body grafts are the thoracic bifurcation and the visceral manifold. The thoracic bifurcation is deployed in the thoracic aorta and provides the proximal seal for the device. For a Type I or II thoracoabdominal aneurysm the proximal seal is in zone 3, for Type III and V the device seals in zone 4. The two limbs of the thoracic bifurcation allows for continued aortic flow while deploying the visceral segment. The visceral manifold is deployed within the larger 20 mm limb of the thoracic bifurcation to set the stage for the visceral debranching. The branches of the visceral manifold extend to the visceral vessel with the use of covered bridging stents and provide distal seal of the manifold. The smaller 16 mm limb of the thoracic bifurcation extends to the infrarenal segment to either seal in zone 9 for a Type I and V and in zone 10 for Type II and III. All other connections in the device make use of sizes that are modular and independent of patient anatomy.

The Medtronic Valiant Thoracoabdominal Stent Graft works to bifurcate aortic flow upstream of the target visceral vessels. This bifurcation has a two-fold benefit. First it allows for aortic flow to be compartmentalized into a visceral segment and an infrarenal segment providing for uninterrupted flow to the visceral vessels as well as the infrarenal segment throughout the procedure. If any of the connections cannot be made or the patient status declines during the procedure, then it can be staged and the connections can be made at a later date. Second, the upstream bifurcation encourages more favorable flow conditions in the bridging stents and target vessels which may prevent target vessel occlusion. This is due to the fact that the bifurcations are upstream providing a sweeping transition into the renal arteries that is smooth providing for relatively laminar flow conditions. The design demonstrates that more central aortic flow is obtained with this design increasing flow rates in the visceral vessels to potentially increase target vessel patency.

The device can be used as an off-the-shelf system, negating the need for lead times associated with custom-built devices. The critical sizing will need to be done with the proximal end of the thoracic bifurcation, distal landing zone in the aorta or iliac arteries, and the bridging stents. The proximal end of the thoracic bifurcation can be sized by choosing any of the available sizes of the Medtronic TAAA thoracic bifurcation stent grafts, and the sizes of the bridging stents can be manipulated by choosing any of the commercially available sizes of the Atrium iCast. The Atrium iCasts are added to the system in-vivo and connected with passive fixation which negates the need to size the main body components based on the target vessel sizes. All other connections in the device make use of sizes that are the same, independent of patient anatomy.

The deployment of this device is also independent of device alignment. Angular alignment of the thoracic bifurcation and the visceral manifold has very little impact on the outcome of the case. Longitudinal alignment is more important, but a safety factor has been built-in by calling for the distal ends of the visceral manifold to be deployed above their target vessels by 1-2 cm. The longitudinal landing should be optimized so that the graft is not landed too low that the connection with the visceral vessels is challenging to make.

Patients included in the study will undergo follow-up at one month, six months, twelve months and then annually for five years.

ELIGIBILITY:
Inclusion Criteria:

1. A patient may be entered into the study if the patient has at least one of the following:

   1. an aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
   2. aneurysm with a history of growth > 0.5 cm in 6 months
   3. saccular aneurysm deemed at significant risk for rupture
   4. symptomatic aneurysm greater than 4.5 cm
2. Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit.
3. Proximal landing zone for the thoracic bifurcation stent graft that has:

   1. ≥ 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA) diameter in the range of 26-42 mm.
   2. adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold.
4. Minimum branch vessel diameter ≥ 5 mm.
5. Iliac artery or aortic distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm.
6. Patient is ≥ 18 years of age.
7. Patient has a life expectancy > 1 year.

Exclusion Criteria:

1. Patient is a good candidate for and elects open surgical repair.
2. Patient can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis.
3. Patient is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site.
4. Patient is unwilling to comply with the follow-up schedule.
5. Patient is unable or refuses to give informed consent.
6. Urgent or emergent presentation.
7. Patient is pregnant or breastfeeding.
8. Patient has a contained rupture.
9. Patient has a ruptured aneurysm.
10. Patient has a dissection in the treated portion of the aorta.
11. Obstructive stenting of any or all of the visceral vessels.
12. Poor performance status including 2 major system failures (cardiovascular, renal, hepatobiliary, neuromuscular).

Medical Exclusion Criteria:

1. Patient has known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
2. Patient has known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed.
3. Patient has an uncorrectable coagulopathy.
4. Patient has a body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment.
5. Patient has had a major surgical or interventional procedure. unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair.
6. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina).
7. Patient has a systemic or local infection that may increase the risk of endovascular graft infection.
8. Baseline creatinine greater than 2.0 mg/dL.
9. History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome).

Anatomical Exclusion Criteria:

1. Thrombus or excessive calcification within the neck of the aneurysm.
2. Anatomy that would not allow maintenance of at least one patent hypogastric artery.
3. Anatomy that would not allow primary or assisted patency of the left subclavian artery.

Expanded Selection Criteria:

Subjects who fail to meet inclusion criteria for the primary study arm may be enrolled under an expanded selection arm if they meet the following criteria.

Inclusion Criteria:

1. Patient that meets the criteria for inclusion in the primary study arm but has one or more of the following criteria which would exclude them from the primary study arm:

   1. Patient has a minimum branch vessel diameter less than 5 mm.
   2. Patients presents urgently or emergently.
   3. Patient has a contained rupture.
   4. Patient has a ruptured aneurysm.
   5. Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated.
   6. Patient has poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular).
   7. Patient's baseline creatinine greater than 2.0 mg/dL.
   8. Patient's anatomy that would not allow for maintenance of at least one hypogastric artery.
   9. Patient's anatomy that would not allow for primary or assisted patency of the left subclavian artery.

   Or
2. Patient that meets the criteria for inclusion in the primary study arm and:

   1. Would not be eligible for the primary study arm per a documented reason other than those outlined above, and
   2. Per the opinion of the Principal Investigator, with concurrence of the IRB, alternative therapies are unsatisfactory and the probable risk of using the investigational device is no greater than the probable risk from the disease or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects free from major adverse events | 30 days
  major adverse events include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke.

SECONDARY OUTCOMES:
Treatment Success at follow-up intervals | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Treatment success includes freedom from: aneurysm enlargement, aneurysm related mortality, aneurysm rupture, conversion to open repair, secondary intervention for migration, Type I and III endoleaks, device integrity failure, and patency related events, renal failure, all-cause mortality, endoleaks, device integrity failure, patency related events and other device related events.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Answini, MD, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No